CLINICAL TRIAL: NCT04287894
Title: A Phase Ib, Open-label, Single-center Study to Assess the Safety of Cancer-immunotherapy Induction With Tremelimumab and Durvalumab Prior to Chemoradiotherapy and/or Resection in the Treatment of Locally Advanced NSCLC.
Brief Title: Assess the Safety of Immunotherapy Induction With Tremelimumab and Durvalumab Prior to Chemoradiotherapy and/or Resection in the Treatment
Acronym: Induction
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on initially defined safety rules not continued with expansion phase of study (too much toxicity with neo-adjuvant immunotherapy)
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N17DTL
Record Dates: First submitted 2019-10-24; First posted 2020-02-27 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Stage III NSCLC
Keywords: No prior radiotherapy to the thorax.; undergoing EBUS and/or mediastinoscopy.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; tremelimumab; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1A (firste cohort) (Experimental): 1 course Durvalumab (1500mg) + Tremelimumab (75mg) + 1 course of Durvalumab (1500mg) followed by CRT
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Pemetrexed; Drug: Cisplatin; Radiation: chemo radiotherapy; Procedure: Resection
- Cohort 2A (Experimental): 2 course Durvalumab (1500mg) + Tremelimumab (75mg) followed by CRT
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Pemetrexed; Drug: Cisplatin; Radiation: chemo radiotherapy; Procedure: Resection
- Cohort 2B (Active Comparator): 2 course Durvalumab (1500mg) + Tremelimumab (75mg) followed by CRT
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Pemetrexed; Drug: Cisplatin; Radiation: chemo radiotherapy; Procedure: Resection

INTERVENTIONS:
Drug: Durvalumab — The IP will be given to the patient as long as there is a clinical benefit, in invertigator's judgment. Per day, 1500 mg
Drug: Tremelimumab — Per day 75mg
Drug: Pemetrexed — 500 mg/m2 on day 1 every 3 weeks for 2 cycles
Drug: Cisplatin — 6 mg / m2 on day 1 every 3 weeks for 2 cycles
Radiation: chemo radiotherapy — Once-daily fraction, 2 Gy per fraction. Total dose is 60 Gy.
Procedure: Resection — After CIT-CRT

SUMMARY:
A Phase Ib, Open-label, Single-center study to assess the safety of cancer-immunotherapy induction with Tremelimumab and Durvalumab prior to Chemoradiotherapy in the treatment of locally advanced NSCLC.

DETAILED DESCRIPTION:
Patients with pathologically proven stage III NSCLC will be treated with CIT-induction. In the feasibility phase, the first cohort (cohort 1A) will receive only 1 course of the immunotherapy doublet followed by a single dose of Durvalumab (Figure 1). The 2nd cohort (Figure 1, cohort 2A) will open for inclusion if 5 to 6 out of 6 patients complete CIT-CRT according to the safety rules (paragraph 6.1.3). In next cohort two courses of Tremelimumab and Durvalumab will be administered. The expansion cohort will be opened (Figure 1, cohort 2B) if this is well tolerated. Patients will be enrolled for cohort 1B in case < 5 out of 6 patients complete CIT-CRT in cohort 2A.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures.

  2. Male or female aged 18 years or older. 3. WHO performance status of 0 or 1. 4. Pathologically proven NSCLC stage III or inoperable stage II (cT1-3N0-1), according to the 8th edition of the AJCC staging, with a clinical indication for concurrent chemo-irradiation. Patients with locoregional recurrent lung tumour following surgery or a second primary cancer are eligible, unless a pneumonectomy was performed.

  5. Patients should be able to receive concurrent chemo radiotherapy treatment as approved by the MDM.

  6. Body weight >30kg 7. Negative pregnancy test (urine or serum) for female patients with childbearing potential; 8. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of ≤ 1% per year, during the treatment period and for at least 180 days after the last dose of Durvalumab and Tremelimumab combination therapy or 1 month after the last dose of chemotherapy, whichever is later.

A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

Examples of contraceptive methods with a failure rate of ≤ 1% per year include bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices (IUDs), and copper IUDs.

The following age-specific requirements apply:

* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

  9. Adequate organ function. Minimum required laboratory data. 10. No major contra-indications for undergoing EBUS and/or mediastinoscopy. 11. For patients included in the two feasibility cohorts a calculation for the mean lung dose (MLD) for radiotherapy will be performed: in both cohorts at least 2 out of 6 patients with a MLD ≥ 16 need to be included.

Exclusion Criteria:

* 1. Patients with grade 3 dyspnoea or worse at baseline (according to CTCAE version 4.03).

  2. Prior radiotherapy to the thorax. 3. Participation in another clinical study with an investigational product during the last 4 weeks.

  4. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study 5. Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of chemotherapy.

  6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.

  7. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

  8. Any condition that, in the opinion of the investigator, would interfere with evaluation of the CRT or interpretation of patient safety or study results.

  9. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with Durvalumab or Tremelimumab may be included only after consultation with the Study Physician.

  10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
  3. Any chronic skin condition that does not require systemic therapy
  4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  5. Patients with celiac disease controlled by diet alone 11. Subject noncompliance that, in the opinion of the investigator or sponsor, warrants withdrawal; eg, refusal to adhere to scheduled visits 12. General contra-indications for immunotherapy:

  <!-- -->

  1. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
  2. Receipt of a live, attenuated vaccine within 30 days prior to enrolment or anticipation that such a live, attenuated vaccine will be required during the study.
  3. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1 or anti-PD-L1 therapeutic antibodies.
  4. Treatment with systemic immunostimulatory agents (including but not limited to interferons or IL-2) within 14 days or five half-lives of the drug (whichever is shorter) prior to enrolment. Current or prior use of immunosuppressive medication within 14 days before the first dose of Durvalumab or Tremelimumab. The following are exceptions to this criterion:

     * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
     * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
     * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
     * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., one-time dose of dexamethasone for nausea) may be enrolled in the study. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.

       13. History of idiopathic pulmonary fibrosis (including bronchiolitis obliterans with organizing pneumonia) or evidence of active pneumonitis on screening chest computed tomography scan.

       14. History of active primary immunodeficiency 15. History of allogeneic transplantation 16. Severe infections within 28 days prior to enrolment, including, but not limited to, hospitalization for complications of infection, bacteraemia, or severe pneumonia or received oral or IV antibiotics within 2 weeks prior to enrolment. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Safety of CIT-induction with Tremelimumab and Durvalumab prior to CRT in stage III NSCLC | 3 months after the last radiation dose.
  Number of patients who complete the multimodality treatment.

SECONDARY OUTCOMES:
the percentage of patients with mediastinal and / or radiological down-staging following CIT-induction allowing a complete resection. | At 7 weeks
Disease free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Overall survival (OS) | From date of randomization until the date of death assessed up to 100 months
1-Year disease control rate (DCR) | week -1 (baseline) until 12 months

CONTACTS AND LOCATIONS:
Overall Officials: W Theelen, MD, Principal Investigator — NKI-AvL
Locations (1):
- Antoni van Leeuwenhoek - Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided